CLINICAL TRIAL: NCT02343562
Title: Probiotics for Prophylaxis of Postoperative Hirschsprungs Associated Enterocolitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Elfiky, MD, Lecturer of Pediatric Surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CAIUNIPEDSURG-CR1; PACTR201408000867421 (Other: PACTR)
Record Dates: First submitted 2015-01-09; First posted 2015-01-22 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Hirschsprung Disease
MeSH Terms: conditions — Hirschsprung Disease | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Probiotic Sachets
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Probiotic Sachets
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotics Group (Active Comparator): Will receive Sachet-form probiotics
  Interventions: Dietary Supplement: Probiotics
- Placebo Group (Placebo Comparator): Will receive off-the-shelf oral multivitamin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics — Probiotics in the form of sachet will be given twice daily for a period of at least 6 months during the trial period.
  Other Names: Lacteol Forte
  Arms: Probiotics Group
Dietary Supplement: Placebo — Multivitamin off-the-counter.
  Other Names: Multisanostol
  Arms: Placebo Group

SUMMARY:
Hirschsprungs Associated Enterocolitis (HAEC) with incidence up to 30% postoperatively. The objective of the trial is to prevent postoperative HAEC by using Probiotics.

DETAILED DESCRIPTION:
Randomised Controlled Study with two arms. All cases following up for post operative Hirschsprungs surgery are included in this study. First arm will receive a probiotics in the form of sachet for 6 months. Second arm will receive a multivitamin as placebo. Comparative analysis between the two groups for baseline and followup prevalence of Hirschsprungs associated enterocolitis.

ELIGIBILITY:
Inclusion Criteria:

* Hirschsprungs disease confirmed preoperative and postoperative specimen pathology

Exclusion Criteria:

* Other cases of Enterocolitis and constipation

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2014-10; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Prevention of Hirschsprung's associated enterocolitis (HAEC) | 6 months
  Absence of HAEC symptoms and signs; absence of fever, abdominal distension, loose stools (diarrhea) , bloody stools during the postoperative period for 6 months.

SECONDARY OUTCOMES:
Improvement of stooling pattern of postoperative Hirschsprung's cases | 6 months
  Bowel habits and motion data are recorded at base line (start of the study) and measured throughout the study. Number of motions per day, stool consistency and periodic culture and sensitivity analysis of the stools. Improvement is measured by optimising stool output to 2-3 times daily, stool consistency according to age should be semi-solid to solids. Stool analysis improvement criteria include better consistency, absence of pus cells or red blood cells and no growth on culture for pathogenic bacteria.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud MA Elfiky, M.D., Principal Investigator — Cairo University
Locations (1):
- Cairo University Pediatric Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] El-Sawaf M, Siddiqui S, Mahmoud M, Drongowski R, Teitelbaum DH. Probiotic prophylaxis after pullthrough for Hirschsprung disease to reduce incidence of enterocolitis: a prospective, randomized, double-blind, placebo-controlled, multicenter trial. J Pediatr Surg. 2013 Jan;48(1):111-7. doi: 10.1016/j.jpedsurg.2012.10.028. PMID 23331802
- [Background] Demehri, Farokh R., et al.